CLINICAL TRIAL: NCT01444118
Title: Phase III, Open-label, Multicentre, Randomised Trial to Establish Safety and Efficacy of an EGF Cancer Vaccine in Inoperable, Late Stage (IIIb/IV) NSCLC Patients Eligible to Receive Standard Treatment and Supportive Care.
Brief Title: A Randomized Trial to Study the Safety and Efficacy of EGF Cancer Vaccination in Late-stage (IIIB/IV) Non-small Cell Lung Cancer Patients
Acronym: NSCLC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The early termination is not related to safety/toxicity but to initiate new Phase III with biomarker to enrich population & to further strengthen OS benefit
Sponsor: Bioven Europe (Industry)
Responsible Party: Sponsor
Organization: Bioven Sdn. Bhd. (Industry)
Masking: None
Other Study IDs: BV-NSCLC-001
Record Dates: First submitted 2011-09-29; First posted 2011-09-30 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EGF Vaccine (Experimental): Patients in this arm will receive a low dose of Cyclophosphamide and the recombinant human rEGF-P64K/Montanide ISA 51 vaccine in addition to Best Supportive Care.
  Interventions: Biological: Therapeutic EGF Vaccine (Cyclophosphamide and the recombinant human rEGF-P64K/Montanide ISA 51 vaccine)
- Best Supportive Care (No Intervention): Patients in this arm will receive best supportive care

INTERVENTIONS:
Biological: Therapeutic EGF Vaccine (Cyclophosphamide and the recombinant human rEGF-P64K/Montanide ISA 51 vaccine) — Patients in this arm will receive a low dose of Cyclophosphamide and the recombinant human rEGF-P64K/Montanide ISA 51 vaccine in addition to Best Supportive Care.
  Arms: EGF Vaccine

SUMMARY:
The vaccine contains humanized recombinant antigen (Epithelial Growth Factor) and an adjuvant. The antibodies induced by vaccination will react with circulating EGF leading to removal of EGF from the circulation. As a result, binding to its target EGF-Receptor is prevented. Blocking of EGF-Receptor is preventing activation and stimulation of proliferation of tumour cell. A Phase III clinical trial on the EGF vaccine is ongoing in Cuba. The result from previous studies demonstrated positive correlation between extended survival and immune response against the vaccination in the late-stage NSCLC patients' age below 60 with improved quality of life. The purpose of this international Phase III trial is to determine whether the recombinant human EGF cancer vaccine is safe, immunogenic and effective in the treatment of stage IIIB/IV NSCLC patients compared to standard treatment and supportive care.

ELIGIBILITY:
Inclusion Criteria:

1. Are aged 20-65 years (inclusive).
2. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
3. Have adequate bone marrow, liver and renal function, as assessed by the Investigator. A sample taken at Screening should confirm that:

   * White blood cell (WBC) count ≥ 3000 per µL
   * Platelet count ≥ 100,000 per µL
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN) (or ≤ 5 x ULN when liver metastases are present)
   * Total bilirubin ≤ 1.5 x ULN
   * Serum creatinine ≤ 1.5 x ULN
4. Have histologically and/or cytologically confirmed diagnosis of NSCLC, corresponding to locally and regionally advanced, inoperable disease (Stage IIIb or Stage IV [as defined by the American Joint Committee on Cancer staging system]), excluding brain metastases.
5. Are eligible to receive first-line chemotherapy (without concurrent thoracic radiotherapy or consolidation radiotherapy).
6. Agree to use double-barrier contraception (males and females alike [if applicable]). A negative pregnancy test must be documented at Screening for females of childbearing potential.

   Note: Females of childbearing potential are defined as those women with less than 2 years after last menstruation and not surgically sterile, while post-menopausal refers to those women with at least 2 years from last menstruation.
7. Have signed a voluntary written informed consent form (ICF). Patients should be cooperative, willing and able to participate and adhere to the Protocol requirements, including their availability for the follow-up.

Exclusion Criteria:

1. Patient has no measurable disease (as defined by RECIST criteria, version 1.1).
2. Patient is a candidate for concurrent chemo-radiotherapy or post chemo thoracic radiotherapy.
3. Patient has a history of known or suspected central nervous system (CNS) metastases.
4. Patient has a history of primary malignancy (except resected non-melanoma skin cancer or curatively treated carcinoma in situ of the cervix), unless in complete remission and off all chemotherapy and/or radiotherapy for that disease for a minimum of 5 years.
5. Patient is taking immunosuppressant drugs such as azathioprine, tacrolimus, cyclosporine, etc. Use is not permitted within 1 month before Screening.
6. Patient is taking any other immunotherapy.
7. Patient has primary or secondary immunodeficiencies (e.g. documented Human Immunodeficiency Virus [HIV]).
8. Patient has autoimmune disease.
9. Patient has undergone splenectomy.
10. Patient is taking oral, intramuscular or intravenous corticosteroids. Use is not permitted within 1 month before Screening. Inhaled corticosteroids to treat respiratory insufficiency (e.g. chronic obstructive pulmonary disease [COPD]), or topical steroids are permitted.
11. Patient has a neurotoxicity (Grade ≥2).
12. Patient has diarrhoea (Grade ≥2).
13. Patient has received other vaccines (with the exception of the influenza vaccine), within 1 month before Screening.
14. Patient has a history of any severe or life-threatening hypersensitivity reaction.
15. Patient has an unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal and metabolic disease).
16. Patient has recent history (within 6 months before Screening) of chronic alcohol or drug abuse which may compromise the patient's safety or ability to participate in study activities.
17. Patient has a history of psychiatric disorder that prevents patients from providing informed consent or following Protocol instructions.
18. Patient is currently enrolled in an investigational device or drug trial, or <1 month since completing an investigational device or drug trial.
19. Female patients who are pregnant or lactating.
20. Patient has any other factor that in the opinion of the Investigator (or designee) would make the patient unsafe or unsuitable for the study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2011-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Each patient will be followed till death occurs within the time frame of study of 3 years

SECONDARY OUTCOMES:
To establish the safety of an EGF cancer vaccine in inoperable, late stage (IIIb/IV) NSCLC patients. | Each patients will be followed till death occurs within the time frame of study of 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Nicolson, Dr., Principal Investigator — Aberdeen Royal Infirmary UK
Locations (1):
- Aberdeen Royal Infirmary, Aberdeen, United Kingdom